CLINICAL TRIAL: NCT03870165
Title: Food First Approach to Stimulate Muscle Protein Synthesis in Healthy Adults
Acronym: Salmon
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Urbana-Champaign (Other)
Responsible Party: Principal Investigator, Nicholas Burd, Assistant Professor, University of Illinois at Urbana-Champaign
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 19293
Record Dates: First submitted 2019-03-08; First posted 2019-03-11 (Actual); Last update posted 2020-09-28 (Actual); Status verified 2020-09

CONDITIONS: Hypertrophy
MeSH Terms: conditions — Hypertrophy | interventions — Resistance Training; Fatty Acids

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Salmon (Active Comparator): After resistance exercise, participants will ingest 3.5 oz of salmon fillet (21g protein, 24g fat) cooked sous-vide.
  Interventions: Behavioral: Resistance exercise; Other: Salmon
- Isolated mixture (Experimental): After resistance exercise, participants will ingest an isolated amino acid and fatty acid mixture matched to the amino acid and fatty acid content of 3.5 oz salmon fillet.
  Interventions: Behavioral: Resistance exercise; Dietary Supplement: Isolated amino acids and fatty acids

INTERVENTIONS:
Behavioral: Resistance exercise — Participants will perform leg press and leg extension immediately prior to ingestion of salmon or isolated mixture
Other: Salmon — Participants will ingest salmon immediately after resistance exercise
  Arms: Salmon
Dietary Supplement: Isolated amino acids and fatty acids — Participants will ingest a mixture of isolated amino acids and fatty acids immediately after resistance exercise
  Arms: Isolated mixture

SUMMARY:
In a crossover design 10 young healthy adults (20-35 y) will receive stable isotope tracer infusions and perform a single bout of resistance exercise. Immediately after exercise participants will ingest either 3.5 oz of Salmon fillet or its constituent macronutrients as isolated amino acids and fat. Repeated blood and breath samples as well as muscle biopsies will be collected to determine whole body amino acid kinetics, muscle amino acid transporters, anabolic signalling and myofibrillar protein synthesis rates during the trials

DETAILED DESCRIPTION:
On both infusion trials, participants will report to the laboratory at 0700 h after an overnight fast. Upon arrival to the lab, the participant will fill out a questionnaire and a baseline breath sample will be collected to determine 13CO2 enrichment by isotope ratio mass spectrometry. A Teflon catheter will be inserted into the antecubital vein for a baseline blood sample (t=-210) and then participants will receive priming doses of NaH13CO2 (2.35 µmol·kg-1), L-[1-13C]leucine (7.6 µmol·kg-1), and L-[ring-2H5]phenylalanine (2.0 µmol·kg-1). Subsequently, a continuous intravenous solution of L-[1-13C]leucine (0.10 µmol·kg-1·min-1) and L-[ring-2H5]phenylalanine (0.05 µmol·kg-1·min-1) will be initiated (t=-210) and maintained over the infusion trials. A second Teflon catheter will be inserted into a heated dorsal vein for repeated arterialized blood sampling and remained patent by a 0.9% saline drip. Breath samples and arterialized blood samples will be collected every 30 to 60 minutes during the postabsorptive and postprandial states. In the post-absorptive state of infusion trial 1, muscle biopsies will be collected at t=-150 and -30 min of infusion to determine basal-state myofibrillar protein synthesis rates, relative skeletal muscle amino acid transporter content, and anabolic-related signaling. In the subsequent cross-over trial only 1 muscle biopsy will be collected at t=-30 for Western blot analysis and postabsorptive myofibrillar protein-bound tracer enrichment. After collection of the resting muscle biopsy at t=-30 for both trials, the participants will perform resistance exercise that consists of 4 sets of 10-12 repetitions or to muscular failure at 65-70% of 1-RM for both leg press and leg extension exercise.

Immediately after the completion of the exercise bout, participants will ingest either 3.5 oz of Salmon fillet or a matched isolated amino acid and fat mixture (t=0). Completion of the meal will mark the start of the postprandial stage and additional muscle biopsies will be collected at t=120 and t=300.

ELIGIBILITY:
Inclusion Criteria:

* Age 20-35 years
* Recreationally-active adults: ≥ 30 min of physical activity at moderate intensity ≥ 3 times per week
* English fluency

Exclusion Criteria:

* Smoking
* Known allergies to fish consumption
* Vegans
* Diagnosed GI tract diseases
* Arthritic conditions
* A history of neuromuscular problems
* Diagnosed cognitive impairments
* Recent (1 year) participation in amino acid tracer studies
* Predisposition to hypertrophic scarring or keloid formation
* Individuals on any medications known to affect protein metabolism (i.e. corticosteroids, non-steroidal anti-inflammatories, or prescription strength acne medications).
* High blood pressure (Systolic > 140 mm HG; Diastolic > 90 mm HG)
* Alcohol consumption >10 drinks per week
* Metabolic disorders (e.g., Metabolic Syndrome, diabetes, thyroid diseases)
* Consumption of thyroid, androgenic or other medications known to affect endocrine function
* Consumption of ergogenic-leves of dietary supplements that may affect muscle mass (e.g., creatine, HMB), insulin-like substances, or anabolic/catabolic pro-hormones (e.g., DHEA) within 6 weeks prior to participation
* Currently pregnant
* A suboptimal diet quality score as assessed by ASA24 dietary records
* Asthma
* Hypogonadism
* Cardiovascular disease, arrhythmias

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-11-22 (Actual); Study Completion 2019-11-22 (Actual)

PRIMARY OUTCOMES:
Fractional synthetic rate of myofibrillar proteins | Postabsorptive for 3 hours, postprandial for 5 hours.
  Myofibrillar protein synthesis rates will be assessed during the postabsorptive period for 3 hr and during the 5 hr after the ingestion of the experimental interventions. This will allow us to assess the change from the postabsorptive to the postprandial period.

SECONDARY OUTCOMES:
Phosphorylation of muscle anabolic signaling | Baseline and at 2 and 5 hours after protein ingestion
  Phosphorylation of anabolic signaling pathways will be assessed in the fasted state and at 2 and 5 hr after the ingestion of the experimental interventions.
Exogenous rate of leucine appearance | 5 hour postprandial phase
  Leucine oxidation rates will be assessed in the fasted state and at multiple time points in the postprandial phase.

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas A Burd, PhD, Principal Investigator — University of Illinois at Urbana-Champaign
Locations (1):
- Freer Hall, Urbana, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Paulussen KJ, Barnes TM, Askow AT, Salvador AF, McKenna CF, Scaroni SE, Fliflet A, Ulanov AV, Li Z, West DW, Bauer LL, Paluska SA, Dilger RN, Moore DR, Boppart MD, Burd NA. Underpinning the Food Matrix Regulation of Postexercise Myofibrillar Protein Synthesis by Comparing Salmon Ingestion With the Sum of Its Isolated Nutrients in Healthy Young Adults. J Nutr. 2023 May;153(5):1359-1372. doi: 10.1016/j.tjnut.2023.02.037. Epub 2023 Mar 2. PMID 36870539